## **Cover Page for Statistical Analysis Plan**

| Sponsor-Investigator: | Catherine R. Olinger |
|-----------------------|-----------------------------------|
| NCT Number: | NCT04272606 |
| Unique Protocol ID: | 201912099 |
| Official Title: | Prospective, Randomized, Double |
| | Blind Study on the Effects of |
| | Tranexamic Acid on Intraoperative |
| | Blood Loss During Lumbar Spinal |
| | Fusion And Instrumentation |
| Date of Document: | 05 December 2023 |

## **Statistical Analysis**

All analyses will be conducted using R statistical software (version 4.3.1). Continuous variables will be summarized using medians and interquartile ranges and comparisons between groups will be done made using Wilcoxon rank sum or Kruskal-Wallis tests. Pairwise analyses within a group will be made using the Wilcoxon signed rank test. Categorical variables will be summarized using counts and percentages, and comparisons between groups will be performed using Pearson  $\chi^2$  test or Fisher exact test. Kendall's tau  $(\tau)$  will be used as a non-parametric test of association between variables. For all analyses, the threshold for significance will be <0.05 without adjustment for multiple comparisons. Variables will be compared between groups by calculating standardized mean differences.